CLINICAL TRIAL: NCT01482091
Title: Intranasal Fentanyl for Initial Treatment of a Vaso-occlusive Crisis: A Randomized, Double Blind Placebo Controlled Trial
Brief Title: Intranasal Fentanyl for Initial Treatment of a Vaso-occlusive Crisis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Marc Fein, Assistant Professor of Pediatrics, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-09-343
Record Dates: First submitted 2011-11-22; First posted 2011-11-30 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Anemia, Sickle Cell; Pain
Keywords: fentanyl; intranasal; sickle cell; vasoocclusive crisis; pain crisis; pediatrics
MeSH Terms: conditions — Anemia, Sickle Cell; Pain; Vaso-Occlusive Crises | interventions — Fentanyl; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Saline (Placebo Comparator)
  Interventions: Drug: Normal Saline
- Intranasal Fentnayl (Experimental)
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Fentanyl Citrate — A single dose of fentanyl citrate (2 mcg/kg; max 100mcg) administered intranasally. Half of the volume will be administered in each nare. The medication will be administered using a mucosal atomization device
  Arms: Intranasal Fentnayl
Drug: Normal Saline — A single dose of equivalent volume of 0.9% Normal Saline will be administered intranasally. Half of the volume will be administered in each nare. The medication will be administered using a mucosal atomization device.
  Arms: Intranasal Saline

SUMMARY:
The purpose of this study is to determine if intranasal fentanyl can decrease the pain of patients with sickle cell disease who present to the pediatric emergency department with a vaso-occlusive crisis.

DETAILED DESCRIPTION:
Principles of therapy for treatment of vaso-occlusive crises include early aggressive analgesic therapy with opiates and non-steroidal anti-inflammatory agents as well as fluid administration. It is known that there is a significant delay in time to administration of analgesics in children with VOC in the ED. The most easily modifiable factor that contributes to delayed opiate administration is route of administration.

Intranasal medication administration is an easy, rapid way to administer opiates with minimal discomfort as well as bypassing first past metabolism and the blood brain barrier. Intranasal fentanyl has been shown to be a safe and effective analgesic for treatment of acute pain in children, reaching therapeutic effect in 2-10 minutes after administration.

The investigators believe that intranasal fentanyl therapy will be able to provide expedited and effective pain therapy to patients with sickle cell disease presenting to the pediatric emergency department with a vaso-occlusive crisis

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease
* Ages 3 years - 21 years

Exclusion Criteria for Enrollment:

* Pregnancy
* Known allergy to Fentanyl
* Usage of daily home opiates

Exclusion Criteria at presentation in ED with a painful crisis:

* Wong Baker FACES Pain Score <6
* Systolic blood pressure < 5 percentile for age
* Oxygen saturation <92% on room air
* Temperature > 102°F
* Respiratory distress
* Priapism
* Isolated abdominal pain
* Isolated headache
* New neurological symptoms
* Severe rhinorrhea or epistaxis
* History of trauma
* Pregnancy

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Fein, MD, Principal Investigator — Children's Hospital at Montefiore; Daniel M Fein, MD, Study Director — Children's Hospital at Montefiore
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were PRE-CONSENTED for the study in the outpatient hematology clinic, inpatient floors prior to discharge or a separate emergency department (ED) visit prior to discharge. This was done to prevent decision making while under emotional duress of a vaso-occlusive crisis (VOC).
  PRE-CONSENT occurred from 12.12.2011-1.8.2015
Pre-assignment Details: 124 subjects were consented for the study. The study drug was only administered one time in the ED if subjects met all inclusion and exclusion criteria when they arrived with a VOC. Only 49 of the 124 consented subjects received the study drug.
Period: Overall Study
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Saline | Intranasal Fentnayl | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (5.1) | 10.6 (5.3) | 11.6 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 19 | 11 | 30
weight [Median (Inter-Quartile Range); unit: kg] | 45 [29 to 70] | 28 [24 to 52.5] | 37 [24.5 to 64]
Type of Sickle Cell Disease [Number; unit: participants] — SS, SC and SB refer to different genotypes of sickle cell disease, commonly referred to as Hemoglobin SS, Hemoglobin SC and Hemoglobin S/Beta thalassemia, respectively
  participants
    SS | 19 | 20 | 39
    SC | 6 | 3 | 9
    SB | 0 | 1 | 1
Duration of VOC [Number; unit: participants]
  <1/2 day | 7 | 9 | 16
  1/2-1day | 5 | 7 | 12
  1-2 day | 6 | 4 | 10
  >2 day | 7 | 4 | 11
Location of VOC [Number; unit: participants]
  Abdomen | 6 | 10 | 16
  Back | 12 | 12 | 24
  Chest | 4 | 7 | 11
  Head | 1 | 4 | 5
  Arms | 5 | 9 | 14
  Legs | 12 | 10 | 22
Oral analgesic within 2h prior to study drug [Number; unit: participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score 20 Minutes After Administration of Study Drug
Description: Change in pain score between 0 and 20 minutes using the Wong Baker FACES pain scale (WBFPS). The WBFPRS has six faces, with each face representing an increasing severity of pain the more rightward it is on the scale (0 is the lowest score , which represents the least amount of pain, while 10 is the highest score which represents the greatest level of pain).. Each face has an even number underneath it, consecutively.
  To calculate the change, the reported pain score at 20 minutes was subtracted from the reported baseline pain score. Thus, the higher change in pain score is indicative of a GREATER change in pain (i.e. greater decrease in pain at 20 minutes compared to baseline). The greatest possible changes in pain would be a 10 (pain score of 10 at baseline and 0 at 20 minutes) representing a DECREASE in pain between the two time points, and -10 (pain score of 0 at baseline and 10 at 20 minutes) representing a INCREASE in pain between the two time points.
Time Frame: Baseline and 20 minutes after administration of study drug
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 24
units on a scale | 1 [0 to 2] | 2 [0.5 to 4]
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Fentnayl; Test type: Superiority or Other; p = 0.048, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Presence of Bradycardia
Description: Number of participants who had bradycardia
Time Frame: Every 5 minutes until 30 minutes after study drug administration
Measure: Number; unit: participants
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 24
participants | 0 | 0

3. Secondary Outcome: Presence of Headache
Time Frame: Participants will be followed for the duration of their ED visit, an expected average of 6 hours
Measure: Number; unit: participants
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 25
participants | 0 | 4
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Fentnayl; Test type: Superiority or Other; p = 0.05, Fisher Exact

4. Secondary Outcome: Admission Rate
Time Frame: This will be assessed at either discharge from the ED or admission to an inpatient unit, an expected average of 6 hours after triage
Measure: Number; unit: participants
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 24
participants | 16 | 13
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Fentnayl; Test type: Superiority or Other; p > 0.05, Chi-squared

5. Secondary Outcome: Length of Stay in ED
Description: Given multiple confounding factors, reliable data was not able to be obtained for this outcome measure
Time Frame: Time from triage until either discharge from the ED or admission to an inpatient unit, an expected average of 6 hours
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Total Amount of Narcotics Administered
Description: Given multiple confounding and extraneous factors, reliable data was not able to be obtained for this outcome measure
Time Frame: Participants will be followed for the duration of their ED visit, an expected average of 6 hours
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Study Drug Administration
Time Frame: Time from triage to adminstration of study drug
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 24 | 25
minutes | 47 (28) | 43 (36)
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Fentnayl; Test type: Superiority or Other; p = 0.68, t-test, 2 sided

8. Secondary Outcome: Change in Pain Score at 10 Minutes
Description: Change in pain score between 0 and 10 minutes using the Wong Baker FACES pain scale (WBFPS). The WBFPRS has six faces, with each face representing an increasing severity of pain the more rightward it is on the scale (0 is the lowest score , which represents the least amount of pain, while 10 is the highest score which represents the greatest level of pain).. Each face has an even number underneath it, consecutively.
  To calculate the change, the reported pain score at 10 minutes was subtracted from the reported baseline pain score. Thus, the higher change in pain score is indicative of a GREATER change in pain (i.e. greater decrease in pain at 10 minutes compared to baseline). The greatest possible changes in pain would be a 10 (pain score of 10 at baseline and 0 at 10 minutes) representing a DECREASE in pain between the two time points, and -10 (pain score of 0 at baseline and 10 at 10 minutes) representing a INCREASE in pain between the two time points.
Time Frame: Baseline and 10 minutes after administration of study drug
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 24
units on a scale | 0 [0 to 2] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Fentnayl; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Pain Score at 30 Minutes
Description: Change in pain score between 0 and 30 minutes using the Wong Baker FACES pain scale (WBFPS). The WBFPRS has six faces, with each face representing an increasing severity of pain the more rightward it is on the scale (0 is the lowest score, which represents the least amount of pain, while 10 is the highest score which represents the greatest level of pain).. Each face has an even number underneath it, consecutively.
  To calculate the change, the reported pain score at 30 minutes was subtracted from the reported baseline pain score. Thus, the higher change in pain score is indicative of a GREATER change in pain (i.e. greater decrease in pain at 30 minutes compared to baseline). The greatest possible changes in pain would be a 10 (pain score of 10 at baseline and 0 at 30 minutes) representing a DECREASE in pain between the two time points, and -10 (pain score of 0 at baseline and 10 at 30 minutes) representing a INCREASE in pain between the two time points.
Time Frame: Baseline and 30 minutes after administration of study drug
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 24
units on a scale | 2 [0 to 2] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Fentnayl; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Pain Score
Description: Due to confounding factors we were unable to obtain reliable data for this outcome
Time Frame: Baseline and immediately prior to IV insertion
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Respiratory Distress
Description: Participants who had respiratory distress within 30 min of study drug administration
Time Frame: Every 5 minutes until 30 minutes after study drug administration
Measure: Number; unit: participants
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 24
participants | 0 | 0

12. Secondary Outcome: Hypotension
Description: Participants who had hypotension within 30 min of study drug administration
Time Frame: Every 5 minutes until 30 minutes after study drug administration
Measure: Number; unit: participants
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 24
participants | 2 | 2

13. Secondary Outcome: Hypoxia
Description: Number of participants who had hypoxia within 30 min of study drug adminsitration
Time Frame: Every 5 minutes until 30 minutes after study drug administration
Measure: Number; unit: participants
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Number analyzed (Participants) | 25 | 24
participants | 0 | 3
Statistical Analysis 1: Comparison: Intranasal Saline vs Intranasal Fentnayl; Test type: Superiority or Other; p > 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Intranasal Saline | Intranasal Fentnayl
Serious Adverse Events (participants affected / at risk) | 2/25 | 5/24
Other Adverse Events (participants affected / at risk) | 9/25 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Saline (N=25) | Intranasal Fentnayl (N=24)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 — No subjects received any intervention for the transient hypoxia
Hypotension (Cardiac disorders) | 2 | 2 — No subjects received any intervention for the transient hypotension
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Saline (N=25) | Intranasal Fentnayl (N=24)
Sleepiness (Nervous system disorders) | 6 | 10
Headache (Nervous system disorders) | 0 | 4
Itching (Skin and subcutaneous tissue disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Nasal Pain (Skin and subcutaneous tissue disorders) | 0 | 3
Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Blood Transfusion (Blood and lymphatic system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No